CLINICAL TRIAL: NCT06722105
Title: Phase I/II Randomized Clinical Trial of Allogeneic Adipose Tissue-derived Mesenchymal Stromal Cells Systemic Infusion in Severe Systemic Sclerosis
Acronym: MSC-AT-SSc
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP211026
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Severe Systemic Sclerosis
Keywords: Systemic autoimmune disease; Allogenic mesenchymal stromal cells infusion
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: Multi-center, three-arm, randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2 infusions of MSC (Experimental)
  Interventions: Biological: 2 infusions of MSC
- 1 infusion of MSC (Experimental)
  Interventions: Biological: 1 infusion of MSC
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: 2 infusions of MSC — 1 MSC(AT) (2x10^6 cells/kg) injection at M0 and 1 MSC(AT) (2x10^6 cells/kg) injection at M3
  Arms: 2 infusions of MSC
Biological: 1 infusion of MSC — 1 MSC(AT) (2x10^6 cells/kg) injection at M0 and 1 placebo injection at M3
  Arms: 1 infusion of MSC
Other: Placebo — Placebo at M0 and M3
  Arms: Placebo

SUMMARY:
Systemic sclerosis (SSc) is a rare, severe and chronic systemic autoimmune disease (AD) characterized by vasculopathy, immune dysregulation and fibrosis leading to multi-organ dysfunction (primarily skin, lungs, heart gastrointestinal tract and kidneys), with high morbidity and mortality, altered health-related quality of life, all at high cost for patients and society.

Treatment are mostly symptomatic and only autologous hematopoietic stem cell transplantation (AHSCT) has shown long term improvement in overall and event-free survival with disease-modifying properties. However, AHSCT is contra-indicated in case of advanced visceral involvement and in eligible patients, it is still associated with risk of toxicity. There is an urgent need to identify safe and effective treatments for severe SSc.

Mesenchymal stromal cells (MSC) are multipotent cells which carry immunomodulatory, pro-angiogenic and anti-fibrotic properties, that can target SSc pathogenesis and its clinical manifestations. The increasing use of MSC, harvested from bone marrow (MSC(M)), adipose tissue (MSC(AT)), or umbilical cord (MSC(UC)) in a variety of indications, provides consistent evidence supporting their safety in humans. The efficacy of MSC(M) intravenous (IV) injection for treating acute graft versus host disease led to their marketing approval in 2012 and MSC(AT) (Alofisel) were approved for severe Crohn's fistula in 2018.

MSC represent a promising therapeutic approach for SSc. We have previously a) shown disease-specific abnormalities in MSC(M) from SSc patients, providing strong rationale to use allogeneic MSC to treat SSc patients, b) published the first phase I/II dose escalation trial using allogenic MSC(M) infusion in 20 severe SSc patients (ClinicalTrials.gov: NCT02213705, PHRC AOM 11-250) with no safety issues, significant improvement in skin fibrosis at 3 to 6 months after infusion which appeared lower thereafter, thereby supporting the need for repeated infusions.

In vitro, experimental and clinical studies suggest that MSC properties vary according to their tissue of origin/source. We demonstrated that compared to MSC(M), MSC(AT) are easier to harvest and display higher proliferative capability before entering senescence, higher genetic stability, and superior immunosuppressive properties.

Considering the above rationale, we hypothesize that use of healthy donors allogeneic MSC(AT) produced by Etablissement Français du Sang (EFS) will demonstrate a) no safety issues, b) an efficacy profile that will increase with repeated infusion of allogeneic MSC(AT) to treat SSc.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent;
2. Willing to comply with all study procedures and be available for the duration of the study;
3. Male or female, aged ≥ 18 and ≤ 70 years of age
4. SSc patients according to American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2013 classification criteria for SSc
5. Severe disease with either:

   * disease duration of 2 years or less with a modified Rodnan skin score (mRss) ≥ 20 and (abnormal CRP > 5 mg/l and/or hemoglobin < 11 g/dL), or
   * mRSS ≥ 15 without any restriction as to disease duration plus at least one major organ involvement as defined by:

     1. respiratory involvement consisting of lung diffusion capacity for carbon monoxide (DLCO) and/or forced vital capacity (FVC) < 80% predicted and evidence of interstitial lung disease : bronchiolar involvement, areas of ground-glass contusions or fibrosis (chest X-ray and/or high resolution computed tomography (HRCT) scan) and/or moderate Pulmonary hypertension with baseline resting systolic pulmonary arterial pressures > 35 mmHg and below 50 mmHg by cardiac echocardiography, or mean pulmonary artery pressure > 20 mmHg and < 40 mm Hg on right heart catheterization;
     2. renal involvement consisting of past renal crisis, microangiopathic hemolytic anemia, and/or renal insufficiency not explained by other causes than SSc;
     3. cardiac involvement consisting of reversible congestive heart failure, atrial or ventricular rhythm disturbances such as recurrent episodes of atrial fibrillation or flutter, recurrent atrial paroxysmal tachycardia, 2nd or 3rd degree AV-block, mild to moderate pericardial effusion and/or presence of MRI involvement (Increased T1 or T2 mapping, late gadolinium enhancement, septal D sign). All causes of organ involvement should be attributed to SSc.
6. Contraindication, inadequate response or unwillingness to undergo AHSCT(determined by patient and physician judgement)
7. Contraindication, inadequate response or unwillingness or adverse events necessitating discontinuation of conventional immunosuppressive therapy (MMF, methotrexate);
8. Women of reproductive potential must use highly effective contraception;
9. Men of reproductive potential must use condoms;
10. Health insurance.

Exclusion Criteria:

1. Age < 18 years and > 70 years
2. Pregnancy or unwillingness to use adequate contraception;
3. Life-threatening end-organ damage defined as: DLCO (corrected for hemoglobin) < 30% predicted; Left ventricular ejection fraction < 40% by cardiac echocardiography; Pulmonary hypertension with baseline resting systolic pulmonary arterial pressures > 50 mmHg by cardiac echocardiography, or mean pulmonary artery pressure > 40 mmHg on right heart catheterization; glomerular filtration rate < 30mL/min
4. Active Hepatitis (ASAT, ALAT > 3 normal)
5. Neoplasms of less than 5 years, except for basal cell or in situ cervix carcinoma or concurrent myelodysplasia,
6. Uncontrolled hypertension
7. Uncontrolled acute or chronic infection
8. HIV-1 or HIV-2 infection
9. Body Mass Index < 16.5 kg/m2
10. Severe psychiatric disorder
11. Bone marrow insufficiency, defined as neutropenia < 1 x 109/L, thrombopenia < 50 x 109/L, anemia < 8 g/dL, lymphopenia < 0,5 x 109/L
12. Inability to provide informed consent
13. Patient included in another interventional clinical trial
14. Patient under tutelle

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment-related Serious Adverse Events | After each infusion
  Defined as Adverse Events (AE) of grade equal or above 3 using the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 classification, at one month after each infusion according to arms (M1, M4) An injection will be considered as not tolerated for any toxicity criteria above grade ≥ 3

SECONDARY OUTCOMES:
Rate of treatment-related Serious Adverse Events (SAE) | At time of infusion
  Adverse Events of grade equal or above 3 CTCAE v5.0 An injection will be considered as not tolerated for any toxicity criteria above grade ≥ 3
Rate of treatment-related Serious Adverse Events (SAE) | Within 24 hours of infusion
  Adverse Events of grade equal or above 3 CTCAE v5.0 An injection will be considered as not tolerated for any toxicity criteria above grade ≥ 3
Rate of treatment-related Serious Adverse Events (SAE) | At 6 months
  Adverse Events of grade equal or above 3 CTCAE v5.0 An injection will be considered as not tolerated for any toxicity criteria above grade ≥ 3
Rate of treatment-related Serious Adverse Events (SAE) | At 9 months
  Adverse Events of grade equal or above 3 CTCAE v5.0 An injection will be considered as not tolerated for any toxicity criteria above grade ≥ 3
Rate of treatment-related Serious Adverse Events (SAE) | At 12 months
  Adverse Events of grade equal or above 3 CTCAE v5.0 An injection will be considered as not tolerated for any toxicity criteria above grade ≥ 3
Mean modified Rodnan skin score (mRSS) difference | Between Month 0 and month 12
  Main efficacy endpoint is assessed by mRSS difference between M0 and M12 Mean modified Rodnan skin score (mRSS) is a semiquantitative score, ranging from 0 (normal) to 3 (severe), used to evaluate the skin thickness in 17 different cutaneous sites (for a total score from 0 to 51). The higher the score, the more severe the disease.
Mean modified Rodnan skin score (mRSS) | At 3 months
  Mean modified Rodnan skin score (mRSS) is a semiquantitative score, ranging from 0 (normal) to 3 (severe), used to evaluate the skin thickness in 17 different cutaneous sites (for a total score from 0 to 51). The higher the score, the more severe the disease.
Mean modified Rodnan skin score (mRSS) | At 6 months
  Mean modified Rodnan skin score (mRSS) is a semiquantitative score, ranging from 0 (normal) to 3 (severe), used to evaluate the skin thickness in 17 different cutaneous sites (for a total score from 0 to 51). The higher the score, the more severe the disease.
WHO performance status | At month 0
  Karnofsky performance scale Score varies betwwen 0 and 5. The lower the score, the less the patient's life is affected.
WHO performance status | At month 3
  Karnofsky performance scale Score varies betwwen 0 and 5. The lower the score, the less the patient's life is affected.
WHO performance status | At month 6
  Karnofsky performance scale Score varies betwwen 0 and 5. The lower the score, the less the patient's life is affected.
WHO performance status | At month 12
  Karnofsky performance scale Score varies betwwen 0 and 5. The lower the score, the less the patient's life is affected.
Scleroderma-Health Assessment Quetionnaire | At month 0
  It determines a disability index (DI), which is calculated as a continuous variable from 0 (no disability) to 3 (severe disability) Steen VA Arthritis et rhumatism 1997 ; 40 : 1984-91
Scleroderma-Health Assessment Quetionnaire | At month 3
  It determines a disability index (DI), which is calculated as a continuous variable from 0 (no disability) to 3 (severe disability) Steen VA Arthritis et rhumatism 1997 ; 40 : 1984-91
Scleroderma-Health Assessment Quetionnaire | At month 6
  It determines a disability index (DI), which is calculated as a continuous variable from 0 (no disability) to 3 (severe disability) Steen VA Arthritis et rhumatism 1997 ; 40 : 1984-91
Scleroderma-Health Assessment Quetionnaire | At month 12
  It determines a disability index (DI), which is calculated as a continuous variable from 0 (no disability) to 3 (severe disability) Steen VA Arthritis et rhumatism 1997 ; 40 : 1984-91
Short Form (36) health survey (SF36v2) | At month 0
  The Short Form (36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
Short Form (36) health survey (SF36v2) | At month 3
  The Short Form (36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
Short Form (36) health survey (SF36v2) | At month 6
  The Short Form (36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
Short Form (36) health survey (SF36v2) | At month 12
  The Short Form (36) Health Survey is a 36-item measure if health status. The score obtained varies between 0 and 100. The higher the score the less disability.
EQ-5D-5L quality of life questionnaire | At month 0
  It evaluates five dimensions : mobility, self-care, usual activities, pain/discomfort and anxiety/depression and each dimension has five levels : no problems, slight problems, moderate problems, severe problems and extreme problems. Answers are given on a 5-point scale by domain, the higher the score, the poorer the quality of life.
EQ-5D-5L quality of life questionnaire | At month 3
  It evaluates five dimensions : mobility, self-care, usual activities, pain/discomfort and anxiety/depression and each dimension has five levels : no problems, slight problems, moderate problems, severe problems and extreme problems. Answers are given on a 5-point scale by domain, the higher the score, the poorer the quality of life.
EQ-5D-5L quality of life questionnaire | At month 6
  It evaluates five dimensions : mobility, self-care, usual activities, pain/discomfort and anxiety/depression and each dimension has five levels : no problems, slight problems, moderate problems, severe problems and extreme problems. Answers are given on a 5-point scale by domain, the higher the score, the poorer the quality of life.
EQ-5D-5L quality of life questionnaire | At month 12
  It evaluates five dimensions : mobility, self-care, usual activities, pain/discomfort and anxiety/depression and each dimension has five levels : no problems, slight problems, moderate problems, severe problems and extreme problems. Answers are given on a 5-point scale by domain, the higher the score, the poorer the quality of life.
Forced Vital Capacity (FVC) | At month 0
Forced Vital Capacity (FVC) | At month 3
Forced Vital Capacity (FVC) | At month 6
Forced Vital Capacity (FVC) | At month 12
Diffusing capacity of Lung for carbon monoxide (DLCO) | At month 0
Diffusing capacity of Lung for carbon monoxide (DLCO) | At month 3
Diffusing capacity of Lung for carbon monoxide (DLCO) | At month 6
Diffusing capacity of Lung for carbon monoxide (DLCO) | At month 12
Response to treatment | At month 3
  Defined as any of the following: decreased mRss > 25%, increased FVC > 10% and/or increased DLCO >10%, without need for further immunosuppression except low dose steroids (below 10mg daily)
Response to treatment | At month 6
  Defined as any of the following: decreased mRss > 25%, increased FVC > 10% and/or increased DLCO >10%, without need for further immunosuppression except low dose steroids (below 10mg daily)
Response to treatment | At month 12
  Defined as any of the following: decreased mRss > 25%, increased FVC > 10% and/or increased DLCO >10%, without need for further immunosuppression except low dose steroids (below 10mg daily)
Progression Free Survival | At month 12
  Defined as the percentage of enrolled patients still alive without evidence of progression 12 months after MSC(AT) injection, with progression defined as any of the following compared to baseline evaluation: decreased FVC > 10% or DLCO > 15%; decrease in LVEF% > 15%; decrease in weight > 15%; decrease in creatinine clearance > 30%; increased mRss > 25% ; and/or increase in SHAQ> 0.5
Global Rank Composite Score (GRCS) | At month 3
  GRCS is based on several outcomes: death, event-free survival (EFS), forced vital capacity (FVC), Health Assessment Questionnaire - Disability Index (HAQ-DI), and Modified Rodnan Skin Score (mRSS). Participants alive ranked higher than those who died; those who survived event-free ranked higher than EFS failures. EFS failure included death, respiratory failure , renal failure , or cardiac failure . The lowest 3 GRCS components are ordinal; improvement, stability, or worsening from baseline.
Global Rank Composite Score (GRCS) | At month 6
  GRCS is based on several outcomes: death, event-free survival (EFS), forced vital capacity (FVC), Health Assessment Questionnaire - Disability Index (HAQ-DI), and Modified Rodnan Skin Score (mRSS). Participants alive ranked higher than those who died; those who survived event-free ranked higher than EFS failures. EFS failure included death, respiratory failure , renal failure , or cardiac failure . The lowest 3 GRCS components are ordinal; improvement, stability, or worsening from baseline.
Global Rank Composite Score (GRCS) | At month 12
  GRCS is based on several outcomes: death, event-free survival (EFS), forced vital capacity (FVC), Health Assessment Questionnaire - Disability Index (HAQ-DI), and Modified Rodnan Skin Score (mRSS). Participants alive ranked higher than those who died; those who survived event-free ranked higher than EFS failures. EFS failure included death, respiratory failure , renal failure , or cardiac failure . The lowest 3 GRCS components are ordinal; improvement, stability, or worsening from baseline.
Composite response index in dcSSc (CRISS) | At month 3
  For early SSc patients only It is a weighted score and includes five measures: modified Rodnan skin score, FVC% predicted, HAQ-DI, patient and clinician global assessments.
  CRISS score is a probability from 0 to 1 that represents the likelihood of a patient achieving overall improvement. The higher the score, the greater the improvement
Composite response index in dcSSc (CRISS) | At month 6
  For early SSc patients only It is a weighted score and includes five measures: modified Rodnan skin score, FVC% predicted, HAQ-DI, patient and clinician global assessments.
  CRISS score is a probability from 0 to 1 that represents the likelihood of a patient achieving overall improvement. The higher the score, the greater the improvement.
Composite response index in dcSSc (CRISS) | At month 12
  For early SSc patients only
Overall survival | At month 12
  For early SSc patients only It is a weighted score and includes five measures: modified Rodnan skin score, FVC% predicted, HAQ-DI, patient and clinician global assessments.
  CRISS score is a probability from 0 to 1 that represents the likelihood of a patient achieving overall improvement. The higher the score, the greater the improvement
Impact of allogeneic MSC(AT) infusion on the immune response | Up to 6 months
  Impact of allogeneic MSC(AT) iv once or twice at 3 months interval on the immune response, including immunophenotyping and alloimmunization up to M6 after starting therapy
Cost effectiveness of the allogeneic MSC(AT) infusion | At month 12
  Once or twice versus no treatment in severe SSc

OTHER OUTCOMES:
Exploring immune landscape in SSc skin biopsies and signatures predicting treatment response | Up to 12 months
  Before and after MSC(AT)
Evaluating new MSC potency assays interrogating MSC efferocytosis | Up to 12 months

IPD SHARING:
Plan to Share IPD: Undecided